CLINICAL TRIAL: NCT00049686
Title: A Phase I Trial Of VNP40101M, A Novel Alkylating Agent, For Patients With Hematologic Malignancies
Brief Title: VNP40101M in Treating Patients With Relapsed or Refractory Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VION-CLI-029; CDR0000258354 (Registry Identifier: PDQ (Physician Data Query)); MDA-DM-02202
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2003-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: acute undifferentiated leukemia; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory anemia with excess blasts; refractory cytopenia with multilineage dysplasia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Chronic; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Leukemia, Hairy Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — laromustine

INTERVENTIONS:
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of VNP40101M in treating patients who have relapsed or refractory leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of VNP40101M in patients with relapsed or refractory leukemia or poor-risk myelodysplastic syndromes.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the antitumor effects of this drug in these patients.

OUTLINE: Patients receive VNP40101M IV over 15 minutes once every 4 weeks.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Relapsed or refractory leukemia for which no standard therapy is anticipated to result in a durable remission OR
* Poor-risk myelodysplastic syndromes

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No uncontrolled arrhythmia
* No uncontrolled congestive heart failure

Other

* No uncontrolled active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed

Chemotherapy

* At least 2 weeks since prior myelosuppressive cytotoxic chemotherapy in the absence of rapidly progressing disease
* At least 48 hours since prior hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy allowed

Surgery

* Not specified

Other

* No other concurrent standard or investigational treatment for leukemia
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States